CLINICAL TRIAL: NCT07033143
Title: Evaluation of the Efficacy and Safety of Adebrelimab Combined With SOX as Adjuvant Therapy for IIIB and IIIC Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-Adjuvant-001
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cance
Keywords: Adjuvant therapy for gastric cancer; Combined immunotherapy; PD-L1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Adebrelimab combined with SOX treatment for 8 cycles, and Adebrelimab maintenance treatment until 1 year
  Interventions: Drug: Adebrelimab+SOX

INTERVENTIONS:
Drug: Adebrelimab+SOX — Adebrelimab: 1200mg, intravenous drip, day 1, 21 days as one cycle, treatment duration is 1 year.
  SOX: Eight cycles after the operation, intravenous infusion of oxaliplatin at 130 mg/m2. On the first day, oral administration of S-1 at 40-60 mg twice a day. From the first to the 14th day, 21 days constitute one cycle.
  Enhanced CT examinations of the chest, abdomen and pelvis were conducted every 9-12 weeks in the first year of treatment. Then have a check-up every 24 weeks.

SUMMARY:
Although the immunotherapy combination regimen has shown good data and safety during the perioperative period of gastric cancer, more clinical studies are still needed to explore the treatment regimens, the number of treatment cycles, the screening of beneficiary populations, and the safety assessment of different drug combinations of immunotherapy combination therapy as adjuvant treatment after gastric cancer surgery.

DETAILED DESCRIPTION:
Although the immunotherapy combination regimen has shown good data and safety during the perioperative period of gastric cancer, more clinical studies are still needed to explore the treatment regimens, the number of treatment cycles, the screening of beneficiary populations, and the safety assessment of different drug combinations of immunotherapy combination therapy as adjuvant treatment after gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old, gender not limited
2. Surgical pathology confirmed as stage IIIB or IIIC gastric cancer or adenocarcinoma of the gastroesophageal junction (AJCC 8th)
3. The patient underwent R0 surgical resection
4. Have an ECOG performance status score of 0 or 1
5. There are available tumor tissues for PD-L1 expression analysis
6. PD-L1 CPS ≥5
7. No liver, peritoneal or distant metastasis, and peritoneal cytology is negative
8. No previous anti-tumor treatments other than surgery, including but not limited to chemotherapy, targeted therapy, and immunotherapy, have been received
9. The patient's physical condition and visceral functions allow for subsequent adjuvant treatments, including chemotherapy, chemoradiotherapy, and PD-L1 inhibitor therapy.
10. The patient's blood routine and biochemical indicators should meet the following standards: Hb≥90g/L, ANC≥1.5*10^9/L, PLT≥100*10^9/L, ALT and AST≤2.5 U/L, TB≤1.5 UNL, and serum creatinine <1 UNL
11. Patients who were willing to follow the treatment plan during the study period
12. Written informed consent must be obtained before enrollment. Patients have the right to withdraw, and subsequent treatment will not be affected.

Exclusion Criteria:

1. Patients with obvious liver metastasis, peritoneal metastasis or distant metastasis;
2. HER2 positive (++/+++);
3. Pregnant or lactating patients;
4. Received previous anti-tumor treatments, including chemotherapy, radiotherapy, targeted therapy or immunotherapy, etc.
5. Have suffered from other malignant tumors in the past 5 years (excluding basal cell or squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ or breast cancer);
6. Uncontrollable pleural effusion, pericardial effusion or ascites;
7. Clinically determined as inoperable or with distant metastasis;
8. Have suffered from severe cardiovascular diseases within 12 months before enrollment, such as symptomatic coronary heart disease, grade ≥II congestive heart failure, uncontrolled arrhythmia, and myocardial infarction;
9. Concurrent upper gastrointestinal obstruction/bleeding or digestive dysfunction or malabsorption syndrome;
10. There was a history of gastrointestinal perforation 6 months before enrollment.
11. Concurrent severe and uncontrolled concurrent infections or other severe and uncontrolled concomitant diseases, moderate or severe renal injury;
12. There are poorly controlled clinical symptoms or diseases of the heart, such as :(1) Grade II or above cardiac insufficiency or echocardiography examination according to the New York Heart Association (NYHA) standards (see Annex 5) :LVEF(left ventricular ejection fraction)<50%; (2) Unstable angina pectoris (3) Myocardial infarction occurred within one year before the start of the study treatment; (4) Supraventricular or ventricular arrhythmias of clinical significance require treatment or intervention; (5)QTc>450ms(male); QTc>470ms(for females)(The QTc interval is calculated using the Fridericia formula; If the QTc is abnormal, three consecutive tests can be conducted at intervals of 2 minutes, and the average value can be taken.
13. Allergic reactions to the drugs used in this study;
14. Immunosuppressive drugs have been used within 4 weeks before the first dose of the study treatment, excluding topical glucocorticoids through nasal spray, inhalation or other routes, or systemic glucocorticoids at physiological doses (i.e., no more than 10mg/ day prednisone or equivalent doses of other glucocorticoids), or hormones used for the prevention of contrast agent allergy;
15. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
16. Those currently accompanied by interstitial pneumonia or interstitial lung disease, or those with a previous history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or other pulmonary fibrosis and organized pneumonia that may interfere with the judgment and management of immune-related pulmonary toxicity (for example, Subjects with oblusive bronchiolitis, pneumoconiosis, drug-associated pneumonia, idiopathic pneumonia, or those with evidence of active pneumonia or severely impaired lung function shown on chest computed tomography (CT) images during the screening period are allowed to have radiation pneumonia and active tuberculosis in the radiation field.
17. There is an active autoimmune disease or a history of autoimmune diseases that may recur (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitinitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects that can be controlled only through hormone replacement therapy can be included]); Subjects with skin diseases that do not require systemic treatment, such as vitiligo, psoriasis, alopecia, controlled type 1 diabetes treated with insulin, or asthma that has been completely relieved in childhood and does not require any intervention in adulthood can be included. Asthma patients who require medical intervention with bronchodilators cannot be included.
18. Use immunosuppressants or systemic hormone therapy within 14 days before the initiation of the study treatment to achieve the purpose of immunosuppression (dose >10mg/ day prednisone or other therapeutic hormones);
19. There was a severe infection within 4 weeks before the initiation of the study treatment, including but not limited to hospitalization due to infection, bacteremia or complications of severe pneumonia; Therapeutic antibiotics were administered orally or intravenously within 2 weeks before the initiation of the study treatment (patients receiving preventive antibiotics (for example, those who are eligible to participate in the study to prevent urinary tract infections or exacerbation of chronic obstructive pulmonary disease);
20. Patients with congenital or acquired immune deficiency (such as HIV-infected individuals);
21. Immunosuppressive drugs have been used within 4 weeks before the first administration;
22. The attenuated live vaccine has been administered within 4 weeks before the first administration or is planned to be administered during the study period;
23. Has received other anti-PD-1 antibody treatments or other immunotherapies targeting PD-1/PD-L1 in the past;
24. Received treatment with other investigational drugs within 28 days before the initiation of the study treatment;
25. Unresolved postoperative complications;
26. According to the researcher's judgment, the patient has other factors that may affect the research results or lead to the forced termination of this study halfway, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, severe laboratory test abnormalities, accompanied by family or social factors, etc., which will affect the patient's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
3-year-DFS rate | up to 3 year
  3-year disease-free survival rate

SECONDARY OUTCOMES:
OS | up to 5 year
  overall survival
AE | up to 5 year
  The incidence rate and grade (including serious adverse events and immune-related adverse events) were determined according to the NCI-CTCAE5.0 criteria

IPD SHARING:
Plan to Share IPD: No